CLINICAL TRIAL: NCT03231228
Title: Phase 4, Open-Label, Single-Dose, Parallel-Group Study to Evaluate the Safety of 1 g of Cefazolin in Pediatric Subjects Weighing 25 to Less Than 60 kg and 2 g of Cefazolin in Pediatric Subjects Weighing at Least 60 kg Scheduled for Surgery
Brief Title: Safety of 1 g and 2 g of Cefazolin in Pediatric Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped with agreement from FDA.
Sponsor: B. Braun Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HC-G-H-1601
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Results first posted 2020-03-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Infection
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Intervention Model Description: Approximately 110 subjects will be enrolled and assigned to 1 of the 2 dose groups in a 1:1 ratio (55 subjects in each group). Subjects with a weight of at least 25 kg but less than 60 kg will receive a single IV dose of 1 g cefazolin. Subjects with a weight of at least 60 kg will receive a single IV dose of 2 g cefazolin. Dose groups will not be balanced by age or gender.
Masking Description: n/a, this is an open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cefazolin 1 g Infusion (Active Comparator): Pediatric surgical subjects weighing at least 25 kg to less than 60 kg will receive a single 30-minute infusion of 1 g cefazolin.
  Interventions: Drug: Cefazolin 1 g Infusion
- Cefazolin 2 g Infusion (Active Comparator): Pediatric surgical subjects weighing at least 60 kg will receive a single 30-minute infusion of 2 g cefazolin.
  Interventions: Drug: Cefazolin 2 g Infusion

INTERVENTIONS:
Drug: Cefazolin 1 g Infusion — 1 g cefazolin infusion for pediatric surgical subjects weighing ≥25 to <60 kg
  Arms: Cefazolin 1 g Infusion
Drug: Cefazolin 2 g Infusion — 2 g cefazolin infusion for pediatric surgical subjects weighing at least 60 kg
  Arms: Cefazolin 2 g Infusion

SUMMARY:
This is a Phase 4, open-label, single-dose, parallel-group, multicenter, safety study of cefazolin (1 g or 2 g) in pediatric subjects between 10 and 17 years of age (inclusive) scheduled for surgery.

DETAILED DESCRIPTION:
Approximately 110 subjects will be enrolled and assigned to 1 of the 2 dose groups in a 1:1 ratio (55 subjects in each group). Subjects with a weight of at least 25 kg but less than 60 kg will receive a single IV dose of 1 g cefazolin. Subjects with a weight of at least 60 kg will receive a single IV dose of 2 g cefazolin. Dose groups will not be balanced by age or gender. Additional subjects may be enrolled if necessary to ensure at least 50 evaluable subjects with complete safety data per dose group complete the study.

In a subset of approximately 40 subjects, 4 PK samples will be obtained to determine the cefazolin plasma concentrations in this population.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is between the ages of 10 and 17 years (inclusive) at the time of giving informed consent.
2. The subject is scheduled for surgery that will last less than 3 hours.
3. The subject and the subject's legally authorized representative voluntarily agree that the subject will participate in this study. In accordance with applicable laws, regulations, and institutional review board requirements, the subject signs or orally agrees to an age-appropriate assent and the subject's legally authorized representative signs both an institutional review board approved informed consent form and Health Insurance Portability and Accountability Act authorization prior to the performance of any screening procedures.
4. For subjects who agree to participate in the PK subgroup additional consent will be obtained.
5. The subject weighs (on Day 1) ≥25 kg but <60 kg for inclusion in 1 g dose group.
6. The subject weighs (on Day 1) ≥60 kg for inclusion in 2 g dose group.
7. The subject has been scheduled for any type of surgery requiring single dose perioperative cefazolin prophylaxis.

Exclusion Criteria:

1. Female subjects who are pregnant or lactating/breastfeeding.
2. Female subjects of childbearing potential who are sexually active and who are not willing to use an effective method of birth control during the study period, eg, oral contraceptives, double barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or have a partner with a vasectomy.
3. The subject has impaired renal function based on the revised Schwartz formula.
4. The subject has a known allergy or hypersensitivity to β lactam/cephalosporin antibiotics, penicillins, corn products, or dextrose containing products or solutions, or any of the other ingredients of Cefazolin for Injection United States Pharmacopeia (USP) and Dextrose Injection USP in DUPLEX.
5. The subject has abnormal vital signs or an abnormal electrocardiograph (ECG) considered by the investigator to be clinically significant.
6. The subject has a result of any laboratory test (or repeat test, if done), obtained as standard of care, that is outside the normal limit of the site's laboratory reference range AND is considered by the investigator to be clinically significant.
7. The subject has a known history of human immunodeficiency virus, hepatitis B, or hepatitis C infection.
8. The subject has a history of alcohol or drug abuse.
9. The subject has received any other investigational drug/device within 30 days prior to the study drug administration.
10. The subject has a history of or is currently smoking or using nicotine-containing substances or electronic cigarettes as determined by medical history or subject's verbal report.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - University of Missouri Health Care System, Columbia, Missouri
  - Children's Medical Center Dallas, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Carilion Clinic, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ancef (cefazolin for injection) [package insert]. GlaxoSmithKline. Research Triangle Park (NC); 2004 [cited 2016 Jun 08] — https://www.accessdata.fda.gov/drugsatfda_docs/label/2004/50461slr139_ancef_lbl.pdf
- See also: Cefazolin and Dextrose for Injection [package insert]. B. Braun Medical Inc. Bethlehem [PA]; revised 10/2015 — https://www.accessdata.fda.gov/drugsatfda_docs/label/2015/050779s025lbl.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cefazolin 1 g Infusion | Cefazolin 2 g Infusion
Started | 33 | 28
Completed | 30 | 28
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefazolin 1 g Infusion | Cefazolin 2 g Infusion | Total
Number analyzed (Participants) | 33 | 28 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 28 | 61
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 17 | 12 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 31 | 24 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 26 | 20 | 46
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 33 | 28 | 61
Weight [Mean (Full Range); unit: kg] | 49.68 [25.9 to 59.3] | 81.49 [60.9 to 122.7] | 64.29 [25.9 to 122.7]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Safety]
Description: Safety will be assessed by monitoring adverse events (AEs), physical examinations, vital signs, ECGs, and clinical laboratory results.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cefazolin 1 g Infusion | Cefazolin 2 g Infusion
Number analyzed (Participants) | 33 | 28
Participants | 13 | 14

2. Secondary Outcome: Cefazolin Plasma Concentration Following Infusion
Description: Concentrations will be determined through analysis of 4 blood samples drawn at 0.5-1, 2, 3, and 4 hours after the start of study drug infusion.
Time Frame: Up to 4 hours after start of study drug infusion
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cefazolin 1 g Infusion | Cefazolin 2 g Infusion
Number analyzed (Participants) | 12 | 11
mcg/mL
  0.5 - 1.0 HR | 124.7 (33.880) | 145.5 (62.116)
  2 HR: number analyzed (Participants) | 11 | 11
  2 HR | 53.51 (14.399) | 93.26 (42.267)
  3 HR: number analyzed (Participants) | 11 | 10
  3 HR | 37.35 (10.273) | 57.74 (24.106)
  4 HR: number analyzed (Participants) | 8 | 9
  4 HR | 27.30 (6.0245) | 45.03 (20.232)

ADVERSE EVENTS:
Time Frame: 39 Days maximum which includes maximum 30 days screening period through 8 days post-study drug administration
Arm/Group | Cefazolin 1 g Infusion | Cefazolin 2 g Infusion
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/28
Other Adverse Events (participants affected / at risk) | 13/33 | 14/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cefazolin 1 g Infusion (N=33) | Cefazolin 2 g Infusion (N=28)
Post-Operative Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cefazolin 1 g Infusion (N=33) | Cefazolin 2 g Infusion (N=28)
Nausea (Gastrointestinal disorders) | 3 | 6
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 1 | 1
Infusion site pain (General disorders) | 2 | 2
Infusion site erythema (General disorders) | 0 | 2
Infusion site warmth (General disorders) | 1 | 1
Catheter site bruise (General disorders) | 1 | 0
Infusion site bruising (General disorders) | 1 | 0
Injection site bruising (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Clumsiness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Incision site pruritus (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site pain (Injury, poisoning and procedural complications) | 1 | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the PI may publish data or results from the Study; provided that the PI submits the proposed publication to Sponsor for review at least sixty (60) days prior to the date of submission to the proposed publication. Sponsor may request that any Confidential Information be removed from the proposed publication other than Study data and results. The Investigator certifies that it shall not publish any Study related material other than per this agreement.

DOCUMENTS (4):
  • Study Protocol (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT03231228/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03231228/SAP_001.pdf
  • Informed Consent Form: Master ICF (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT03231228/ICF_002.pdf
  • Informed Consent Form: PK Master ICF (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT03231228/ICF_003.pdf